CLINICAL TRIAL: NCT05829694
Title: Health Outcomes of Parents With Cystic Fibrosis (HOPeCF): A Retrospective Analysis of Impact of Parenthood on Lung Function
Brief Title: Health Outcomes of Parents With Cystic Fibrosis
Acronym: HOPeCF
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Traci Kazmerski, Assistant Professor of Pediatrics, University of Pittsburgh
Other Study IDs: STUDY22010135; 1R01HL161164-01A1 (NIH); KAZMER22A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2023-03-08; First posted 2023-04-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis; Parenthood Status
Keywords: cystic fibrosis; parenthood; highly-effective modulator therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: Individuals diagnosed with cystic fibrosis who became a first-time parent between January 1, 2012 and December 31, 2022.
  Interventions: Other: Parental Status
- Non-parents: Individuals diagnosed with cystic fibrosis who have never been a parent.

INTERVENTIONS:
Other: Parental Status — The aim of the study is to assess the impact parenthood has on health outcomes.
  Groups: Parents

SUMMARY:
This project will determine the health impact of parenthood on people with cystic fibrosis (CF). The study team will use retrospective data to provide relatively immediate evidence on parenthood's effect on pulmonary health.

DETAILED DESCRIPTION:
This co-funded study sponsored by the National Institutes of Health and the CF Foundation (CFF) will seek to determine the health impact of parenthood on people with CF in the era of CF transmembrane conductance regulator (CFTR) modulators. To provide relatively immediate evidence on parenthood's effect on pulmonary health and the influence of the introduction and use of all available CFTR modulators, in Aim 1 the study team will assess changes in pre- vs. intra-parenthood percent predicted forced expiratory volume in 1 second (ppFEV1) in a retrospective longitudinal cohort study linking CFF patient registry (CFFPR) data with cross-sectional surveys collected from 249 new parents attending participating United States CF centers between 2012-2022. The study team will identify predictors and timing of lung function loss using 747 non-parents from participating centers as a comparison group and examine the impact of CFTR modulators on parental health.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CF diagnosis with sweat or genotype analysis
* Participant in the CFFPR
* Became a first-time parent between the years 2012-2022 (exposure arm only)

Exclusion Criteria:

* Lung transplant prior to becoming a first-time parent (exposure arm) or prior to study period (control)
* Does not speak/read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cystic fibrosis who are participants in the Cystic Fibrosis Foundation's Patient Registry.
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
FEV1 | 2012-2022
  Rate of decline of ppFEV1 as reported in the CFFPR

SECONDARY OUTCOMES:
Rate of pulmonary exacerbations | 2012-2022
  Rate of pulmonary exacerbations as reported in the CFFPR
Rate of hospitalizations | 2012-2022
  Rate of hospitalizations as reported in the CFFPR
Clinic visit attendance | 2012-2022
  Clinic visit attendance as reported in the CFFPR
BMI | 2012-2022
  BMI as reported in the CFFPR
Medication Use | 2012-2022
  Medication use as reported in the CFFPR
CFRD Control | 2012-2022
  HbgA1c as reported in the CFFPR
Microbiologic profile | 2012-2022
  Presence of specific types of bacteria, mycobacteria, fungus in cultures as reported in the CFFPR

CONTACTS AND LOCATIONS:
Overall Officials: Traci M Kazmerski, MD, MS, Principal Investigator — University of Pittsburgh
Locations (8):
- United States (8):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - UPMC, Pittsburgh, Pennsylvania
  - University of Texas-Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No